CLINICAL TRIAL: NCT05677347
Title: A Randomized, Double-blind, Placebo Controlled, Single and Repeat Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of Inhaled GSK3923868 in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Phase 1, Single and Repeat Dose Study to Assess Safety, Tolerability, and Pharmacokinetics (PK) of GSK3923868 in Participants With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 214075
Record Dates: First submitted 2023-01-09; First posted 2023-01-10 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: Single ascending dose; Repeat dose; Phosphatidylinositol 4-kinase beta (PI4KB) inhibitor; Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Intervention Model Description: The same cohort of participants will move from Part 1 (single ascending doses treatment periods 1 and 2) to Part 2 (repeat dose treatment period 3)
Who Masked: Participant, Investigator
Masking Description: The participants and investigators will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD (Experimental): Eligible participants will receive a single dose (SD) of GSK3923868 500 microgram (mcg) in Treatment Period 1 followed by a single dose of placebo matching GSK3923868 in Treatment Period 2. Participants will also receive a repeat dose (RD) of GSK3923868 1500 mcg in Treatment Period 3. There will be a washout period between each treatment period. Participants will have a follow-up of 14 days after the last dose of GSK3923868.
  Interventions: Drug: GSK3923868; Drug: Placebo
- GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD (Experimental): Eligible participants will receive a single dose of GSK3923868 500 mcg in Treatment Period 1 followed by a single dose of GSK3923868 1000 mcg in Treatment Period 2. Participants will also receive a repeat dose of placebo matching GSK3923868 in Treatment Period 3. There will be a washout period between each treatment period. Participants will have a follow-up of 14 days after the last dose of GSK3923868.
  Interventions: Drug: GSK3923868; Drug: Placebo
- GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD (Experimental): Eligible participants will receive a single dose of GSK3923868 500 mcg in Treatment Period 1 followed by a single dose of GSK3923868 1000 mcg in Treatment Period 2. Participants will also receive repeat dose of GSK3923868 1500 mcg in Treatment Period 3. There will be a washout period between each treatment period. Participants will have a follow-up of 14 days after the last dose of GSK3923868.
  Interventions: Drug: GSK3923868
- Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD (Experimental): Eligible participants will receive a single dose of placebo matching GSK3923868 in Treatment Period 1 followed by a single dose of GSK3923868 1000 mcg in Treatment Period 2. Participants will also receive a repeat dose of GSK3923868 1500 mcg in Treatment Period 3. There will be a washout period between each treatment period. Participants will have a follow-up of 14 days after the last dose of GSK3923868.
  Interventions: Drug: GSK3923868; Drug: Placebo

INTERVENTIONS:
Drug: GSK3923868 — GSK3923868 will be administered
Drug: Placebo — Placebo will be administered
  Arms: GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD; GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD; Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD

SUMMARY:
This is a two parts study, a single ascending dose followed by 14-days repeat dosing. The single ascending dose part will assess two dose levels of GSK3923868 or placebo across two treatment periods 1 and 2 in a single cohort of participants with a washout period of a minimum of 5 days after each treatment periods. The repeat dose part will assess repeated one dose level of GSK3923868 or placebo in treatment period 3 with up to 14 days of follow up in the same cohort of participants. The duration of study participation for treatment period 1, 2 and 3 will be 6, 6 and up to 29 days (including follow up), respectively.

ELIGIBILITY:
Inclusion Criteria:

* Between 40 and 70 years of age.
* Confirmed diagnosis of COPD for greater than (>) 6 months.
* Participant is a smoker or an ex-smoker with a smoking history of at least 10 pack years.
* A female participant is eligible to participate if she is not pregnant or breastfeeding and agrees to use contraceptives during the study (for women of childbearing potential only).

Exclusion Criteria:

* Participant has poorly controlled or unstable COPD.
* Participant has a past or current medical condition(s) or disease(s) that is/are not well controlled.
* Participant has had a respiratory tract infection treated with antibiotics within 4 weeks prior to screening.
* Participant requires regular treatment with oral corticosteroids or has received a course of oral or parenteral corticosteroids within 4 weeks prior to screening.
* Participant requires long-term oxygen therapy.
* Current enrolment or past participation in a clinical trial within 30 days before this study starts.
* Positive tests for human immunodeficiency virus (HIV), hepatitis B and C, or Coronavirus disease-19 (COVID-19).
* Positive pre-study drug (except for as results of opioids prescribed for medical reasons and/or inadvertent consumption of poppy seeds) /alcohol screening result.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, a key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All the 12 participants were enrolled and randomized in the study.
Groups:
- GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD: Eligible participants received a single dose (SD) of GSK3923868 500 microgram (mcg) in Treatment Period 1 followed by a single dose of placebo matching GSK3923868 in Treatment Period 2. Participants also received a repeat dose (RD) of GSK3923868 1500 mcg in Treatment Period 3. There was a washout period between each treatment period. Participants had a follow-up of 14 days after the last dose of GSK3923868.
- GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD: Eligible participants received a single dose of GSK3923868 500 mcg in Treatment Period 1 followed by GSK3923868 1000 mcg in Treatment Period 2. Participants also received a repeat dose of placebo matching GSK3923868 in Treatment Period 3. There was a washout period between each treatment period. Participants had a follow-up of 14 days after the last dose of GSK3923868.
- GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD: Eligible participants received a single dose of GSK3923868 500 mcg in Treatment Period 1 followed by GSK3923868 1000 mcg in Treatment Period 2. Participants also received repeat dose of GSK3923868 1500 mcg in Treatment Period 3. There was a washout period between each treatment period. Participants had a follow-up of 14 days after the last dose of GSK3923868.
- Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD: Eligible participants received a single dose of placebo matching GSK3923868 in Treatment Period 1 followed by GSK3923868 1000 mcg in Treatment Period 2. Participants also received a repeat dose of GSK3923868 1500 mcg in Treatment Period 3. There was a washout period between each treatment period. Participants had a follow-up of 14 days after the last dose of GSK3923868.
Period: Treatment Period 1 (3 Days)
Arm/Group | GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 1 (up to 6 Days)
Arm/Group | GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (3 Days)
Arm/Group | GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Washout Period 2 (up to 6 Days)
Arm/Group | GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 3 (up to 15 Days)
Arm/Group | GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD
Started | 3 | 3 | 3 | 3
Completed | 3 | 3 | 3 | 3
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | GSK3923868 500 mcg SD/Placebo SD/GSK3923868 1500 mcg RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/Placebo RD | GSK3923868 500 mcg SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Placebo SD/GSK3923868 1000 mcg SD/GSK3923868 1500 mcg RD | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 67.7 (2.31) | 59.3 (5.69) | 63.3 (7.23) | 68.0 (1.00) | 64.6 (5.50)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Gender categories (with 0<n<11) are combined into one 'De-identified' category to maintain participant confidentiality and privacy, as they could lead to participant re-identification.
  Participants
    De-identified | 3 | 3 | 3 | 3 | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race categories (with 0<n<11) are combined into one 'De-identified' category to maintain participant confidentiality and privacy, as they could lead to participant re-identification.
  Participants
    De-identified | 3 | 3 | 3 | 3 | 12

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs) Following Single Dose of GSK3923868
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. An SAE is any untoward medical occurrence that, at any dose: results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect or any other situation according to medical or scientific judgment. Adverse events which were not serious, were considered as non-serious adverse events.
Time Frame: Up to 18 days
Population: This analysis was performed on Safety Population which included all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo SD: Participants received single dose of placebo matching GSK3923868 in Treatment Periods 1 and 2.
- GSK3923868 500 mcg SD: Participants received single dose of GSK3923868 500 mcg in Treatment Period 1.
- GSK3923868 1000 mcg SD: Participants received single dose of GSK3923868 1000 mcg in Treatment Period 2.
Arm/Group | Placebo SD | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Non-SAE | 1 | 2 | 1
  SAE | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Non-SAEs and SAEs Following Repeat Dose of GSK3923868
Description: as for outcome 1
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Groups:
- Placebo RD: Participants received repeat dose of placebo matching GSK3923868 in Treatment Period 3.
- GSK3923868 1500 mcg RD: Participants received repeat dose of GSK3923868 1500 mcg in Treatment Period 3.
Arm/Group | Placebo RD | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 3 | 9
Participants
  Non-SAE | 2 | 4
  SAE | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology and Clinical Chemistry Laboratory Parameters Following Single Dose of GSK3923868
Description: The laboratory measurements included hematology and clinical chemistry. The parameters evaluated were Basophil, Eosinophil, Erythrocyte Mean Corpuscular Hemoglobin, Erythrocyte Mean Corpuscular Volume, Erythrocytes, Hematocrit, Hemoglobin, Lymphocyte, Monocyte, Neutrophils, Platelets and Reticulocytes, Alanine Aminotransferase, Albumin, Alkaline phosphatase, Aspartate Aminotransferase, Bilirubin, Calcium, Creatinine, Direct Bilirubin, Glucose, Potassium, Sodium and Urea. Number of participants with clinically significant changes in hematology and clinical chemistry and were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 18 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SD | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Hematology | 0 | 0 | 0
  Clinical Chemistry | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Changes in Hematology and Clinical Chemistry Laboratory Parameters Following Repeat Dose of GSK3923868
Description: as for outcome 3
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo RD | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 3 | 9
Participants
  Hematology | 0 | 0
  Clinical Chemistry | 0 | 0

5. Primary Outcome: Number of Participants With Clinically Significant Changes in Urinalysis Parameters Following Repeat Dose of GSK3923868
Description: Urine samples were collected at indicated time points for the analysis of urinalysis parameters including specific gravity, potential of hydrogen (pH) of urine, presence of glucose, protein, erythrocytes, ketones, bilirubin, urobilinogen, nitrite, leukocyte esterase in urine by dipstick. Number of participants with clinically significant changes in urinalysis parameters were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo RD | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 3 | 9
Participants | 0 | 0

6. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs and 12-lead Electrocardiogram (ECG) Findings Following Single Dose of GSK3923868
Description: Vital signs included systolic and diastolic blood pressure, pulse rate and respiratory rate were measured with the participant in semi-supine position after at least 10 minutes rest. Tympanic Temperature was also measured as a vital sign but did not require positioning or rest prior to measuring. Twelve-lead electrocardiogram were performed in a semi-supine position after at least 10 minutes rest using an ECG machine that automatically calculates the heart rate and measures PR interval, QRS duration, QT and corrected QT intervals (QTc) intervals. Number of participants with clinically significant changes in vital signs and ECG parameters were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 18 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SD | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 6 | 9 | 9
Participants
  Vital Signs | 0 | 0 | 0
  12-Lead ECG | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Clinically Significant Changes in Vital Signs and 12-lead Electrocardiogram (ECG) Findings Following Repeat Dose of GSK3923868
Description: as for outcome 6
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo RD | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 3 | 9
Participants
  Vital Signs | 0 | 0
  12-Lead ECG | 0 | 0

8. Primary Outcome: Number of Participants With Clinically Significant Changes in Spirometry Measurements Following Single Dose of GSK3923868
Description: Spirometry included forced expiratory volume in 1 second (FEV1) for lung function assessment. FEV1 is an important measure of pulmonary function and is the maximum amount of air that can be forced out in one second after taking a deep breath. Spirometry assessments were performed in triplicate with the highest value reported. Number of participants with clinically significant changes in spirometry measurements were reported. Clinical significance was determined by the investigator.
Time Frame: Up to 18 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo SD | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 6 | 9 | 9
Participants | 0 | 0 | 0

9. Primary Outcome: Number of Participants With Clinically Significant Changes in Spirometry Measurements Following Repeat Dose of GSK3923868
Description: as for outcome 8
Time Frame: Up to 29 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo RD | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 3 | 9
Participants | 0 | 0

10. Secondary Outcome: Area Under the Plasma-concentration Time Curve From Time Zero (Pre-dose) to 24 Hours (AUC [0-24]) of GSK3923868 for Single Dose
Description: Blood samples were collected at the indicated time points for pharmacokinetic (PK) analysis of GSK3923868. Pharmacokinetic analysis was conducted using standard non-compartmental method with WinNonlin.
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6, 24 hours post-dose on Day 1 in Treatment Periods 1 and 2
Population: This analysis was performed on Pharmacokinetic (PK) Population which included all randomized participants in the Safety Population who had at least 1 dose of GSK3923868 and at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* picograms per milliliter
Arm/Group | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 9 | 9
Hours* picograms per milliliter | 23463.81 (24.02) | 46553.52 (21.29)

11. Secondary Outcome: Area Under the Plasma-concentration Time Curve From Time Zero (Pre-dose) to Time of the Last Quantifiable Concentration (AUC[0-t]) of GSK3923868 for Single Dose
Description: Blood samples were collected at the indicated time points for PK analysis of GSK3923868. Area under the concentration-time curve from time zero to the time of the last quantifiable concentration values were reported.
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6, 24 hours post-dose on Day 1 in Treatment Periods 1 and 2
Population: This analysis was performed on PK Population which included all randomized participants in the Safety Population who had at least 1 dose of GSK3923868 and at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were considered as non-missing values).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* picograms per milliliter
Arm/Group | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 9 | 9
Hours* picograms per milliliter | 23443.19 (23.96) | 46519.91 (21.28)

12. Secondary Outcome: Area Under the Plasma-concentration Time Curve From Time Zero (Pre-dose) to 6 Hours (AUC [0-6]) of GSK3923868 for Repeat Dose
Description: as for outcome 10
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6 hours post-dose on Day 1 and Day 14 in Treatment Period 3
Population: This analysis was performed on PK Population which included all randomized participants in Safety Population who had at least 1 dose of GSK3923868 and at least 1 non-missing PK assessment (Non-quantifiable [NQ] values were considered as non-missing values). Only those participants who were measured and analyzed (i.e., contributed data reported in table) were included in 'Overall Number of Participants Analyzed' field. 'Number Analyzed' signifies participants evaluable for specified time points.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hours* picograms per milliliter
Groups:
- GSK3923868 1500 mcg RD: Participants received repeat dose of GSK3923868 1500 mcg (500 mcg*3) in Treatment Period 3.
Arm/Group | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 9
Hours* picograms per milliliter
  Day 1 | 42593.74 (19.93)
  Day 14: number analyzed (Participants) | 8
  Day 14 | 40787.96 (12.96)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of GSK3923868 for Single Dose
Description: as for outcome 10
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6, 24 hours post-dose on Day 1 in Treatment Periods 1 and 2
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 9 | 9
Picograms per milliliter | 4823.19 (26.72) | 10042.80 (11.93)

14. Secondary Outcome: Time to Reach Cmax (Tmax) of GSK3923868 for Single Dose
Description: Blood samples were collected at the indicated time points for analysis of tmax of GSK3923868. The tmax was obtained directly from the concentration-time data. The tmax was analyzed with the non-compartmental methods with WinNonlin.
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6, 24 hours post-dose on Day 1 in Treatment Periods 1 and 2
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD
Number analyzed (Participants) | 9 | 9
Hours | 1.00 [0.8 to 2.0] | 1.00 [0.8 to 2.0]

15. Secondary Outcome: Cmax of GSK3923868 for Repeat Dose
Description: as for outcome 10
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6 hours post-dose on Day 1 and Day 14 in Treatment Period 3
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Picograms per milliliter
Arm/Group | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 9
Picograms per milliliter
  Day 1 | 14081.13 (13.69)
  Day 14 | 13854.60 (25.57)

16. Secondary Outcome: Tmax of GSK3923868 for Repeat Dose
Description: as for outcome 14
Time Frame: Pre-dose and 5, 15, 30, 45 minutes, 1, 2, 4, 6 hours post-dose on Day 1 and Day 14 in Treatment Period 3
Population: as for outcome 11
Measure: Median (Full Range); unit: Hours
Arm/Group | GSK3923868 1500 mcg RD
Number analyzed (Participants) | 9
Hours
  Day 1 | 0.95 [0.8 to 2.0]
  Day 14 | 1.00 [0.8 to 2.0]

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected up to 18 days for single dose cohorts and up to 29 days for repeat dose cohorts
Description: All-cause mortality, SAEs and Non-SAEs were reported for the Safety Population which included all participants who received at least 1 dose of study treatment. AEs were reported treatment-wise.
Arm/Group | Placebo SD | GSK3923868 500 mcg SD | GSK3923868 1000 mcg SD | Placebo RD | GSK3923868 1500 mcg RD
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/9 | 0/9 | 0/3 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/9 | 0/9 | 0/3 | 0/9
Other Adverse Events (participants affected / at risk) | 1/6 | 2/9 | 1/9 | 2/3 | 4/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo SD (N=6) | GSK3923868 500 mcg SD (N=9) | GSK3923868 1000 mcg SD (N=9) | Placebo RD (N=3) | GSK3923868 1500 mcg RD (N=9)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Taste disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT05677347/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT05677347/SAP_001.pdf